CLINICAL TRIAL: NCT01584583
Title: Blood Pressure Monitor Clinical Test (Cuff Range: 22 Cm-36cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AndonHealth6
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Blood Pressure
Keywords: BP

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- blood pressure monitor: Cuff circumference:22cm-36cm
- stethoscopy: Cuff circumference: 22cm-36cm

SUMMARY:
The purpose of this study is to monitor the blood pressure level of the patient using a preformed cuff ranged 22 cm-36 cm.

ELIGIBILITY:
Inclusion Criteria:

* cuff circumference: 22cm-36cm

Exclusion Criteria:

Ages: 24 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resident of a community
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2012-02; Study Completion 2012-04 (Actual)